CLINICAL TRIAL: NCT01247987
Title: Comparison of Transfers of Thawed Blastocysts Versus Blastocysts Derived From Thawed Bipronuclear Oocytes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruce Shapiro M.D. (Industry)
Responsible Party: Sponsor-Investigator, Bruce Shapiro M.D., Medica Director, Fertility Center of Las Vegas
Organization: Fertility Center of Las Vegas (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAIRB 10-0018
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
Keywords: IVF, assisted reproduction, embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blastocyst cryopreservation (Active Comparator): Subjects randomly assigned to this arm of the study will have all of their embryos cryopreserved at the blastocyst stage, followed by thaw and transfer in a subsequent menstrual cycle.
  Interventions: Procedure: Blastocyst cryopreservation
- Bipronuclear oocyte cryopreservation (Experimental): Subjects randomly assigned to this arm of the study will have all of their bipronuclear oocytes cryopreserved, followed by thaw, extended culture, and transfer in a subsequent menstrual cycle.
  Interventions: Procedure: Bipronuclear oocyte cryopreservation

INTERVENTIONS:
Procedure: Blastocyst cryopreservation — Embryos cryopreserved at the blastocyst stage
  Arms: Blastocyst cryopreservation
Procedure: Bipronuclear oocyte cryopreservation — Bipronuclear oocyte cryopreservation.
  Arms: Bipronuclear oocyte cryopreservation

SUMMARY:
The purpose of this study is to determine if cryopreservation at the blastocyst stage followed by embryo thaw and transfer is as effective as cryopreservation of bipronuclear oocytes followed by post-thaw extended culture (PTEC), and blastocyst transfer. Effectiveness will be measured by the rate of ongoing pregnancy at 10 weeks gestation.

DETAILED DESCRIPTION:
Subjects will be randomized to one of two study groups during their cycles of in vitro fertilization (IVF). In one group, the subjects will have all of their embryos cryopreserved at the blastocyst stage, followed by thaw and transfer in a subsequent cycle. In the other group, subjects will have all of their embryos cryopreserved at the bipronuclear oocyte stage, followed by thaw, extended culture, and transfer in a subsequent cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient seeking autologous in vitro fertilization (IVF) treatment.
2. Cycle day 3 serum concentration of follicle stimulating hormone (FSH) less than 10.0 IU/l.
3. Baseline total antral follicle count observed on ultrasound with at least eight antral follicles.
4. 18 to 40 years of age.
5. Ability to read and understand English.

Exclusion Criteria:

1. Embryo biopsy (a.k.a. pre-implantation genetic diagnosis (PGD)).
2. Any condition that, in the opinion of the physician or principal investigator, would place the patient at undue risk under this protocol or would otherwise make the protocol inappropriate for that subject.
3. No minors will be enrolled in this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 10 weeks gestation
  Ultrasonically confirmed fetal heart motion at 10 weeks gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Center of Las Vegas, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C. Freeze-all at the blastocyst or bipronuclear stage: a randomized clinical trial. Fertil Steril. 2015 Nov;104(5):1138-44. doi: 10.1016/j.fertnstert.2015.07.1141. Epub 2015 Aug 5. PMID 26255088